## Effect Of Probiotic Supplementation on The Immune System in Patients with Ulcerative Colitis in Amman, Jordan

By

## Lana Mustafa Agraib

Supervisor

Dr. Mohammed Isam Yamani

Co-Supervisor

Dr. Reema Fayez Tayyem

Funded by the University of Jordan

**22 November 2023** 

NCT04223479

## **Statistical Analysis**

Statistical analyses were performed using Statistical Package for Social Science (IBM® SPSS® Statistics; Version 21.0, version for Windows, 2019, USA). Mean and standard deviation (SD) were calculated for the continuous variables. Frequencies and percentages were used to describe categorical variables. The frequency of participants in terms of categorical variables was compared using the X² test. To check the normal distribution of continuous variables, the Shapiro-Wilk test was applied. Independent samples T-test was used to detect differences between placebo and probiotics groups in terms of continuous variables. A paired t-test was used to assess withingroup changes in biochemical parameters (IgG, IgM, IgA, IL-1, IL-6, IL10, TNF-α, and CRP) from baseline to the end of the study. A p-value < 0.05 was considered statistically significant. All outcomes were calculated by intention-to-treat (ITT) and perprotocol (PP) analyses. For ITT analysis, all randomized patients who took at least one tablet of study medication were included. For PP analysis all protocol violators (patients' dropout or loss of follow-up) were excluded.